CLINICAL TRIAL: NCT03245723
Title: Cardiac Function and Metabolism in Young Adults Born Premature
Brief Title: Cardiac Function and Metabolism in Young Adults Born Premature (PET-MRI)
Acronym: PET-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-0238; UL1TR000427 (NIH); A534285 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*P (Other: UW Madison); Protocol Version 4/23/2019 (Other: UW Madison)
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Infant,Premature
Keywords: premature adults; premature; premature lung function; premature cardiac function; MRI; PET
MeSH Terms: conditions — Premature Birth | interventions — Respiratory Physiological Phenomena; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Young adults born premature (some of them are registered on the National Lung Project) and Healthy Controls will undergo pulmonary function testing, cardiac positron emission tomography, and cardiac magnetic resonance imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm (Active Comparator): Participants born premature either registered on the National Lung Project (currently in their late twenties) or not registered on the National Lung Project Cohort (current age ranges 18-35 years).
  All the participants in this group will undergo Pulmonary Function Testing, Electrocardiogram, Positron Emission Tomography, and Magnetic Resonance Imaging.
  Interventions: Procedure: Pulmonary Function Testing; Procedure: Electrocardiogram; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging
- Term - Healthy Controls (Placebo Comparator): Healthy individuals that were not born premature. Individuals are ages 18-35. Subjects will undergo Pulmonary Function Testing, Electrocardiogram, Positron Emission Tomography, and Magnetic Resonance Imaging.
  Interventions: Procedure: Pulmonary Function Testing; Procedure: Electrocardiogram; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Pulmonary Function Testing — Subjects will undergo Spirometry and Plethysmography
Procedure: Electrocardiogram — Subjects will undergo an electrocardiogram to ensure sinus rhythm
Procedure: Positron Emission Tomography — Subjects will undergo positron emission tomography to detect images of the heart
Procedure: Magnetic Resonance Imaging — Subjects will undergo positron magnetic resonance imaging to detect images of the heart

SUMMARY:
The purpose of this research is to determine the effect of premature birth on later heart function and metabolism.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of premature birth on cardiac function, cardiac metabolism, and oxidative stress in a cohort of young adults born prematurely using cardiac positron emission tomography/magnetic resonance imaging and mitochondrial respiration studies.

ELIGIBILITY:
Inclusion Criteria:

* National Lung Project Cohort only- birth weight <1500g and a gestational age <36 weeks
* Adults born preterm (Non-National Lung Project) only- gestational age ≤32 weeks OR birth weight ≤ 3lbs 5oz
* Healthy Controls only- No personal history of known cardiovascular or pulmonary disease

Exclusion Criteria:

* Metabolic Disorders that would affect Fludeoxyglucose uptake
* Contraindications to positron emission tomography and/or magnetic resonance imaging
* Pregnancy, if a female of child-bearing potential
* A personal history of Type I or Type II diabetes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara N Goss, MD, Principal Investigator — The University of Wisconsin School of Medicine and Public Health
Locations (1):
- UW Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 52 enrolled participants, no data was collected for 2 participants due to COVID. 50 participants were allocated to intervention.
Groups:
- Preterm: Participants born premature either registered on the National Lung Project (currently in their late twenties) or not registered on the National Lung Project Cohort (current age ranges 18-35 years).
  All the participants in this group will undergo Pulmonary Function Testing, Electrocardiogram, Positron Emission Tomography, and Magnetic Resonance Imaging.
  Pulmonary Function Testing: Subjects will undergo Spirometry and Plethysmography
  Electrocardiogram: Subjects will undergo an electrocardiogram to ensure sinus rhythm
  Positron Emission Tomography: Subjects will undergo positron emission tomography to detect images of the heart
  Magnetic Resonance Imaging: Subjects will undergo positron magnetic resonance imaging to detect images of the heart
Period: Overall Study
Arm/Group | Preterm | Term - Healthy Controls
Started | 32 | 18
Completed | 27 | 17
Not Completed | 5 | 1
Not completed — Bigeminy precluding hypoxia exposure | 1 | 0
Not completed — Claustrophobia from wearing the mask | 1 | 0
Not completed — Having to abruptly stop the scan to use the restroom | 2 | 0
Not completed — Image acquisition/reconstruction failure | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preterm | Term - Healthy Controls | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Current age of participants
  years | 26.1 (4.2) | 25.4 (4.0) | 25.75 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 10 | 33
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 31 | 16 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 30 | 16 | 46
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Gestational age (Neonatal Characteristics) [Mean (Standard Deviation); unit: Weeks] — Neonatal characteristics-gestational age of participants at the time of birth
  Weeks | 29.2 (2.5) | 39.8 (1.0) | 34.5 (1.75)
Birth weight (Neonatal Characteristics) [Mean (Standard Deviation); unit: Grams] | 1225 (397) | 3397 (572) | 2311 (484.5)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Glucose Uptake During Normoxic Rest (µg/Min)
Description: Cardiac glucose uptake will be measured via 18F-fluorodeoxyglucose (FDG) PET-MRI.
Time Frame: Visit 1 (1 day)
Population: Data was not collected for 4 preterm participants due to following reasons:
  * bigeminy precluding hypoxia exposure (N=1),
  * claustrophobia from wearing the mask (N=1),
  * having to abruptly stop the scan to use the restroom (N=2).
Measure: Mean (Standard Deviation); unit: µg/min
Arm/Group | Preterm | Term - Healthy Controls
Number analyzed (Participants) | 28 | 18
µg/min | 0.689 (0.546) | 0.540 (0.454)
Statistical Analysis 1: Comparison: Preterm vs Term - Healthy Controls; Test type: Other — Descriptive statistics; p = 0.38, Wilcoxon Rank Sum test

2. Primary Outcome: Change in Glucose Uptake From Normoxia to Hypoxia (µg/Min)
Description: Cardiac glucose uptake will be measured via 18F-fluorodeoxyglucose (FDG) PET-MRI.
Time Frame: Visit 1 (1 day)
Population: 5 preterm and 1 term participants did nor receive the allocated intervention due to :
  * bigeminy precluding hypoxia exposure (N=1 preterm),
  * claustrophobia from wearing the mask (N=1 preterm),
  * having to abruptly stop the scan to use the restroom (N=2 preterm).
  * image acquisition/reconstruction failure (n = 2,1 preterm and 1 term)
Measure: Mean (Standard Deviation); unit: µg/min
Arm/Group | Preterm | Term - Healthy Controls
Number analyzed (Participants) | 27 | 17
µg/min | -0.264 (0.588) | -0.003 (0.390)
Statistical Analysis 1: Comparison: Preterm vs Term - Healthy Controls; Test type: Other — Descriptive statistics; p = 0.12, Wilcoxon Rank Sum test

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Preterm | Term - Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/18
Other Adverse Events (participants affected / at risk) | 0/32 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03245723/Prot_SAP_003.pdf